CLINICAL TRIAL: NCT03182413
Title: Therapeutic Impact of THN102 on Attention, Wakefulness and Cognitive Performance During Total Sleep Deprivation in Healthy Subjects
Brief Title: Impact of THN102 on Attention, Wakefulness and Cognitive Performance During Total Sleep Deprivation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theranexus (Industry)
Collaborators: Institut de recherche biomédicale des armées (IRBA), Bretigny sur Orge, France (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THN102-102
Record Dates: First submitted 2017-06-06; First posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Sleep Deprivation
Keywords: modafinil; connexin; sleep deprivation; cognitive performance
MeSH Terms: conditions — Sleep Deprivation | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- PBO (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- MOD (Active Comparator): Modafinil 100mg
  Interventions: Drug: Modafinil
- THN102 100/1 (Experimental): modafinil 100 mg + 1 mg flecainide
  Interventions: Drug: THN102
- THN102 100/3 (Experimental): modafinil 100 mg + 3 mg flecainide
  Interventions: Drug: THN102
- THN102 100/9 (Experimental): modafinil 100 mg + 9 mg flecainide
  Interventions: Drug: THN102

INTERVENTIONS:
Drug: Placebo
  Arms: PBO
Drug: Modafinil
  Arms: MOD
Drug: THN102
  Arms: THN102 100/1; THN102 100/3; THN102 100/9

SUMMARY:
Study Objectives: THN102 is a new combination between modafinil and flecainide low-dose, a documented glial connexin inhibitor. Efficacy of THN102 was compared to modafinil and to placebo on parameters impaired by total sleep deprivation (SD, lasting 40h).

Methods: 20 healthy male subjects participated in a double-blind, randomised, incomplete-block 3-period cross-over trial involving 5 treatments (n=12 per group): placebo (PBO), modafinil 100 mg (MOD), and combinations THN102 (modafinil 100 mg and 1, 3 or 9 mg flecainide as THN1, THN3 and THN9), as 3 oral doses over 18h.

ELIGIBILITY:
Main inclusion Criteria:

1. Male subjects considered healthy and aged between 18 and 40 years
2. Subject with a body mass index (BMI) between 18 and 30 kg/m2

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Sustained attention (PVT) | 5 hours post treatment
  Mean speed at the 10 min Psychomotor vigilance test (PVT)

SECONDARY OUTCOMES:
Sustained attention (PVT) AUC | AUC of PVT speed during TSD
  AUC of speed values at the 10 min Psychomotor vigilance test (PVT)
Mental flexibility | 16,5 hours post treatment
  Wisconsin card sorting test
Mental inhibition | 16,5 hours post treatment
  GO-noGO
Working memory | 16,5 hours post treatment
  2-Back

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Sauvet, MD, PhD, Principal Investigator — Institut de Recherche Biomedicale des Armees; Françoise Brunner-Ferber, PhD, Study Director — Brunner Naga

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Duchene A, Perier M, Zhao Y, Liu X, Thomasson J, Chauveau F, Pierard C, Lagarde D, Picoli C, Jeanson T, Mouthon F, Dauvilliers Y, Giaume C, Lin JS, Charveriat M. Impact of Astroglial Connexins on Modafinil Pharmacological Properties. Sleep. 2016 Jun 1;39(6):1283-92. doi: 10.5665/sleep.5854. PMID 27091533
- [Derived] Sauvet F, Erblang M, Gomez-Merino D, Rabat A, Guillard M, Dubourdieu D, Lefloch H, Drogou C, Van Beers P, Bougard C, Bourrrilhon C, Arnal P, Rein W, Mouthon F, Brunner-Ferber F, Leger D, Dauvilliers Y, Chennaoui M, Charveriat M. Efficacy of THN102 (a combination of modafinil and flecainide) on vigilance and cognition during 40-hour total sleep deprivation in healthy subjects: Glial connexins as a therapeutic target. Br J Clin Pharmacol. 2019 Nov;85(11):2623-2633. doi: 10.1111/bcp.14098. Epub 2019 Sep 15. PMID 31419329
- See also: Related Info — http://www.theranexus.com